CLINICAL TRIAL: NCT03216616
Title: Guided Self-Management Intervention Targeting Fatigue in Rheumatic Inflammatory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Extrastiftelsen (Other); Norsk revmatikerforbund (Unknown)
Responsible Party: Principal Investigator, Elin Fjerstad, Psychologist, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/395 (REK)
Record Dates: First submitted 2017-07-05; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Fatigue; Inflammatory Rheumatism
Keywords: fatigue; Inflammatory Rheumatism; Coping; self-efficacy
MeSH Terms: conditions — Fatigue; Rheumatic Fever | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with inflammatory rheumatic diseases (Experimental): The patients will participate in a cognitive behavioural therapy intervention
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy

SUMMARY:
Fatigue is common and debilitating in rheumatic inflammatory diseases as for other chronical medical conditions. The purpose of this study is to develope and evaluate a cognitive behavioural intervention targeting fatigue. The aim of the intervention is to improve fatigue self-management by changing behavioral and cognitive factors contributing to perceived fatigue. Levels of fatigue, depressive symptoms and self esteem will be measured before, after and three months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

• Men and women over 18 years with inflammatory rheumatic diseases and fatigue at Department of Rheumatology, Diakonhjemmet Hospital

Exclusion Criteria:

* Unable to provide informed consent
* Unable to read and understand Norwegian
* Unable to complete a survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Screening of the perceived level of fatigue in patients with inflammatory rheumatic disease | 2-10 minutes
  Patients with rheumatic inflammatory diseases suffering from fatigue will be asked to complete the Chalder Fatigue Questionnaire
Screening of depressive symptoms in patients with inflammatory rheumatic disease and fatigue | 2-10 minutes
  Patients with rheumatic inflammatory diseases suffering from fatigue will be asked to complete the Patient Health Questionnaire-9 (PHQ-9)
Screening of the patients perceived self efficacy in coping with fatigue | 10-15 minutes
  The patients will be asked to answer questions about fatigue, activity and rest, sleep problems, worrying and rumination.
Reduce perceived fatigue and increase perceived self efficacy in relation to coping with fatigue in patients with inflammatory rheumatic diseases | 6 weeks-6 months
  Patients enrolled in the study will attend a course or an individual treatment with a clinical psychologist aimed to reduce symptoms of fatigue and improve their self efficacy by means of Cognitive Behaviour Therapy (CBT)
Detection of changes in perceived levels of fatigue | 2-10 minutes
  Patients will be asked to complete the Chalder Fatigue Questionnaire one month and three months after receiving CBT. Results will be compared to the scores obtained prior to CBT.
Detection of changes in symptoms of depression | 2-10 minutes
  The patients will be asked to complete the Patient Health Questionnaire-9 (PHQ-9) one month and three months after receiving CBT. Results will be compared to the scores obtained prior to CBT.
Detection of changes in the patients perceived self efficacy in coping with fatigue | 10-15 minutes
  The patients will be asked to answer questions about fatigue, activity and rest, sleep problems, worrying and rumination one month and three months after receiving CBT. Results will be compared to the scores obtained prior to CBT.

IPD SHARING:
Plan to Share IPD: No